CLINICAL TRIAL: NCT04391946
Title: National Prospective and Retrospective Follow-up of Patients With COVID-19 Infected Chronic Lymphocytic Leukemia / Lymphocytic Lymphoma or Waldenström Disease
Brief Title: Observatory of Patients With Chronic Lymphocytic Leukemia / Lymphocytic Lymphoma or Waldenstrom Disease Infected With COVID-19
Acronym: COVID19_LLC-MW
Status: Completed | Type: Observational
Sponsor: French Innovative Leukemia Organisation (Other)
Collaborators: Institut de cancérologie Strasbourg Europe (Other)
Responsible Party: Sponsor
Other Study IDs: FILO-COVID19_LLC-MW
Record Dates: First submitted 2020-05-13; First posted 2020-05-18 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Chronic Lymphocytic Leukemia, Lymphocytic Lymphoma or Waldenstrom Disease
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Routinely Collected Health Data

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Data registry — Collection of clinical data, treatment regimens and survival data

SUMMARY:
The COVID-19 epidemic (Coronavirus Disease 2019) which is currently raging in France is an emerging infectious disease linked to a virus of the genus coronavirus (SARS-CoV-2). The first cases were reported in Wuhan, China, in late December 2019 [1]. Globally, it has been placed in the "pandemic" stage by the WHO since March 11, 2020. Coronavirus viruses have been responsible for epidemics in the past such as the SARS epidemic in 2002 (Syndrome Severe Acute Respiratory) linked to the SARS-CoV virus, or the epidemic of MERS (Middle East Respiratory Syndrome) that affected the Middle East in 2012.

Patients with chronic lymphocytic leukemia (CLL) / lymphocytic lymphoma or Waldenstrom Disease (WD) therefore represent a population at high risk of developing a severe form in the event of COVID-19 infection.

To date, no data is available in the literature to assess the impact of the COVID-19 epidemic in this population of patients with CLL / lymphocytic lymphoma or WD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic lymphocytic leukemia / lymphocytic lymphoma or Waldenstrom disease according to the criteria of the WHO 2016 with a proven or probable infection by COVID-19 according to the following criteria:
* Proven infection: PCR positive regardless of the radio-clinical picture (Other tests made available later and having good diagnostic performance will be accepted)
* Probable infection: the diagnosis of probable infection is retained in case of negative PCR or not made if presence of at least 2 major criteria or of a major criterion associated with at least 2 minor criteria among the following, in the absence other documented cause.
* Major criteria:

  * Fever
  * Loss of smell / taste
  * At least one respiratory sign among cough, dyspnea, chest pain
  * Radiological signs suggestive of the scanner (areas or diffuse appearance of frosted glass, condensations including pseudonodular condensations, association of frosted glass and condensation within the same lesion, nodules and micronodules, thickening of the interlobular septa) or on an X-ray of the thorax ( interstitial, alveolo-interstitial or alveolar syndrome, unilateral or bilateral)
  * Notion of storytelling with a person whose SARS-CoV-2 infection has been formally documented
* Minor criteria

  * Aches
  * Sore throat
  * Rhinorrhea
  * Headache
  * Diarrhea
  * Abdominal pain
  * Frank asthenia
  * Conjunctivitis

Exclusion Criteria:

* Patient opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 infected patients with chronic lymphocytic leukemia / lymphocytic lymphoma or Waldenström disease
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2020-03-14 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Prognostic factors for healing of COVID-19 infection | Day 0
  Hematological pathology Description

SECONDARY OUTCOMES:
Medical care of Coronavirus infection | within 12 months after diagnosis
  Describe the management carried out concerning Coronavirus infection and its impact on the treatment of hemopathy.
national epidemiological monitoring | through study completion, an average of 2 years
  Allow national epidemiological monitoring and regularly inform the hematology community.

CONTACTS AND LOCATIONS:
Overall Officials: Luc-Matthieu FORNECKER, Pr, Principal Investigator — French Innovative Leukemia Organisation
Locations (22):
- France (22):
  - Chu Angers, Angers
  - CHU Jean Minjoz - Hématologie, Besançon
  - Hôpital Avicenne - Centre de Recherche Clinique, Bobigny
  - CHU Estaing - Hématologie Clinique Adulte, Clermont-Ferrand
  - Chu Creteil, Créteil
  - CHU Grenoble - Hématologie, Grenoble
  - Chd Vendee, La Roche-sur-Yon
  - Centre Hospitalier du Mans, Le Mans
  - Hôpital Saint Vicent de Paul, Lille
  - Centre Léon Bérard - Hématologie, Lyon
  - Institut Paoli Calmette, Marseille
  - Hopital E.Muller, Mulhouse
  - CHU DE NANTES - Hematologie clinique, Nantes
  - Hopital Pitie Salpetriere Service Hematologie Clinique - Pavillon de L'Enfant Et Adolescent, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hôpital de la Milétrie - Hématologie et Thérapie Cellulaire, Poitiers
  - Hôpital Robert Debré - Hématologie Clinique, Reims
  - Centre Henri Becquerel - Service Hématologie Clinique, Rouen
  - Hôpital Hautepierre - Hématologie, Strasbourg
  - IUCT ONCOPOLE - Hématologie, Toulouse
  - Hôpital Bretonneau - Hématologie et Thérapie Cellulaire, Tours
  - CHU Nancy Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No